CLINICAL TRIAL: NCT07247812
Title: The Effects of Transcutaneous Spinal Cord Stimulation on Upper Extremity Function in Children and Young People With Hemiplegic Cerebral Palsy
Brief Title: tSCS in Children and Young People With HCP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Professor Sarah Astill, Professor, University of Leeds
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024-NCT59
Record Dates: First submitted 2025-10-02; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy Spastic Hemiplegic
Keywords: Cerebral palsy; Transcutaneous Spinal Cord Stimulation; Hemiplegic Cerebral Palsy; Upper Extremity Function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous spinal cord stimulation (tSCS) combined with Upper Limb Training Task (ULTT) (Experimental): One session will involve transcutaneous spinal cord stimulation (tSCS) combined with ULTT
  Interventions: Device: Digimer DS8R
- ULTT ONLY (No Intervention): one session with ULTT only (no stimulation; tSCS)

INTERVENTIONS:
Device: Digimer DS8R — Transtcuatne Electrical stimulation will be delivered using the Digimer DS8R. The tSCS will be administered in one session only, during which participants will receive continuous tSCS simultaneously with Upper Limb Motor Training (ULTT).
  Arms: transcutaneous spinal cord stimulation (tSCS) combined with Upper Limb Training Task (ULTT)

SUMMARY:
This work will examine if a technique called Transcutaneous Spinal cord stimulation (tSCS), when used with concurrent specific arm and hand exercises, helps improve arm and hand movements in CYP with HCP.

Does Transcutaneous Spinal Cord Stimulation (tSCS), when combined with specific arm and hand exercises, improve upper limb function in children and young people (CYP) with Hemiplegic Cerebral Palsy (HCP)?

-To determine the feasibility and effectiveness of Transcutaneous Spinal Cord Stimulation (tSCS) combined with targeted arm and hand exercises in improving the upper limb function in children and young people with Hemiplegic Cerebral Palsy (HCP).

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a condition that affects movement and posture due to brain development issues in babies or young children. Hemiplegic CP (HCP) is a condition where one side of the body is paralysed. Symptoms like stiffness in the arms and legs usually appear early and can make everyday tasks, such as reaching or holding objects difficult. Improving arm and hand function is crucial for increasing independence and quality of life for children with HCP. This study investigates a technique called Transcutaneous Spinal Cord Stimulation (tSCS). tSCS uses sticky pads placed on the skin to deliver a mild electrical current. This current stimulates nerves to help them send signals to the muscles, potentially improving arm and hand movements. Research has demonstrated that tSCS can provide benefits in the lower limb for children and young people (CYP) with CP, those with spinal cord injuries and healthy individuals. In this project, we will test the feasibility and effectiveness of tSCS in 18 CYP (aged 12-21 years) with HCP. The participant will attend two sessions. Each session will last approximately 60-90 minutes and will include:

* A Baseline Assessment (before training)
* A 30-minute Upper Limb Task Training (ULTT)
* One session will involve transcutaneous spinal cord stimulation (tSCS) combined with ULTT
* One session will involve ULTT only (no stimulation)
* The order is randomised, meaning participants do the stimulation session first or second
* A Post-Training Assessment

ELIGIBILITY:
Inclusion Criteria

* Age and Gender: Boys and girls aged 12 to 21 years.
* Diagnosis: Are diagnosed with Hemiplegic Cerebral Palsy (HCP).
* Hand Function: Are experiencing difficulties with hand functions in daily activities.
* Medical Stability: Have stable medical conditions without cardiopulmonary disease or seizures.
* Motor Capability: Are capable of performing simple motor tasks such as reaching, touching, or grasping objects.
* Availability: Are able to attend two sessions
* Consent informed: Are able to provide informed consent (or if under 16, will need to have a parent or legal guardian who is willing to provide consent on their behalf).
* Language: Are able to speak English (and if under 16, their parent or legal guardian must also be able to speak English)

Exclusion Criteria

* Other Neurological Conditions: Have neurological diseases other than cerebral palsy.
* Blood Pressure: Have uncontrolled or high blood pressure.
* Recent Surgeries: Have recently undergone significant surgeries (neurological, cardiac, respiratory, or metabolic) without sufficient recovery time.
* Severe Diseases: Have cardiovascular or pulmonary diseases.
* Medical Complications: Have ongoing medical complications such as unhealed fractures, contractures, or active infections or cancer.
* Protocol Compliance: Are unable to follow study protocols safely.
* Epilepsy History: Have a personal or family history of epilepsy.
* Recent Injections: Have had botulinum toxin injections within the past six months.
* Implanted Devices: Have implanted devices like pacemakers or baclofen pumps.
* Exclusion of Participants with Recent Research Involvement: Participants who have taken part in any clinical research study within the last 3 months will be excluded.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Participants with stimulation-site skin reaction (Yes/No; photographic assessment) | At the first session: Baseline (pre-tSCS) and immediately post-tSCS
  Standardised photographs of the back will be obtained at each time point and reviewed by an independent clinician (not part of the study team). A skin reaction is defined as any visible erythema at/near the electrode site and will be recorded on a Yes/No erythema scale (0 = No erythema; 1 = Yes erythema). Results will be reported as the number and proportion of participants with ≥1 skin reaction during the session and by time point.
Heart Rate Category (beats per minute) | [Time Frame: Baseline (pre-tSCS); During tSCS (10 minutes after start); Immediately post-tSCS (within 10 minutes after end) during a single session.
  Heart rate will be measured immediately before and after tSCS using an OMRON M3 device. For each participant, a blinded independent clinician will classify the post-stimulation change relative to Baseline as one of three categories: Increased, Decreased, or No Apparent Change. Study results will be summarised as the number and proportion of participants in each category and described narratively.
Hand Strength Index (dynamometry) | Session 1[first visit]: Pre (Baseline, before tSCS); Session 1 [first visit]: Post (immediately after tSCS, within 10 minutes); Session 2 [second visit]: Pre (Baseline, before tSCS); Session 2 [sv]: Post (immediately after tSCS, within 10 minutes)
  Handgrip and pinch strength will be measured with handheld dynamometers (adjustable handle/pads; peak-hold). At each time point, participants perform 3 maximal attempts per measure; the average (mean) is calculated for handgrip and for pinch. Results will be summarised as mean (SD) by timepoint and change from pre to post within each session (Post - Pre). Component means (handgrip and pinch) will be presented descriptively as supportive information.
Jebsen-Taylor Hand Function Test total time (seconds) | Session 1[first visit]: Pre (Baseline, before tSCS); Session 1 [first visit]: Post (immediately after tSCS, within 10 minutes); Session 2 [second visit]: Pre (Baseline, before tSCS); Session 2 [sv]: Post (immediately after tSCS, within 10 minutes)
  Hand function will be assessed with the Jebsen-Taylor Hand Function Test (JTHFT). The protocol includes three subtests: (1) picking up small common objects; (2) stacking checkers; (3) lifting large light and large heavy cans (~1 lb). Each subtest is timed to completion. Testing is administered with the less affected hand first, then the more affected hand; the primary outcome is the Total Score for the more affected hand. Results will be summarised as mean (SD) seconds by timepoint and change from pre to post within each session (Post - Pre). (Scores for the less affected hand may be presented descriptively as supportive data.)
Muscle Activity: Mean motor threshold to elicit ≥50 µV sEMG response (mA) - Delsys Trigno / Digitimer DS8R | Session 1: Pre (Baseline, before tSCS); Session 1: Post (immediately after tSCS, within 10 minutes); Session 2: Pre (Baseline, before tSCS); Session 2: Post (immediately after tSCS, within 10 minutes).
  Muscle activity will be assessed with surface EMG (Delsys Trigno). Sensors will be placed on the more affected arm over the abductor pollicis brevis, flexor carpi radialis, and extensor carpi radialis longus. Single spinal pulses (1 ms biphasic square-wave) will be delivered every ~5 s using a Digitimer DS8R. For each muscle at each time point, the motor threshold is defined as the lowest stimulation amplitude (mA) that produces an evoked sEMG response ≥50 µV. The participant-level outcome is the mean motor threshold (mA) across the three muscles. Results will be summarised as mean (SD) mA by timepoint and change from Baseline to Post.
Modified Ashworth Scale (0-4; higher = worse) - worst upper-limb muscle score (more affected limb) | Session 1[first visit]: Pre (Baseline, before tSCS); Session 1 [first visit]: Post (immediately after tSCS, within 10 minutes); Session 2 [second visit]: Pre (Baseline, before tSCS); Session 2 [sv]: Post (immediately after tSCS, within 10 minutes)
  Spasticity will be assessed with the Modified Ashworth Scale (MAS), scored 0, 1, 1+, 2, 3, 4 (0 = no increase in tone; 4 = rigid; higher scores indicate worse spasticity). The following muscles on the more affected upper limb will be tested in a fixed order: elbow flexors, wrist flexors, finger flexors. At each timepoint, the primary outcome is the worst (highest) MAS score across the tested muscles. Results will be summarised as median by timepoint and change from Pre to Post within each session (Post - Pre).
Systolic Blood Pressure Category (mmHg) | Baseline (pre-tSCS); During tSCS (10 minutes after start); Immediately post-tSCS (within 10 minutes after end) during a single session.
  Systolic blood pressure will be measured immediately before and after tSCS using an OMRON M3 device. For each participant, a blinded independent clinician will classify the post-stimulation change relative to Baseline as one of three categories: Increased, Decreased, or No Apparent Change. Study results will be summarised as the number and proportion of participants in each category and described narratively.
Diastolic Blood Pressure Category (mmHg) | Baseline (pre-tSCS); During tSCS (10 minutes after start); Immediately post-tSCS (within 10 minutes after end) during a single session.
  Diastolic blood pressure will be measured immediately before and after tSCS using an OMRON M3 device. For each participant, a blinded independent clinician will classify the post-stimulation change relative to Baseline as one of three categories: Increased, Decreased, or No Apparent Change. Study results will be summarised as the number and proportion of participants in each category and described narratively.

SECONDARY OUTCOMES:
Participant-reported experience with stimulation - response frequencies (project-specific questionnaire) | Immediately post-final tSCS session [first session] (within 10 minutes), single administration.
  A project-specific Participant Feedback Questionnaire (PFQ-tSCS), completed by the participant or caregiver, will capture experience with stimulation across predefined domains: comfort, ease of participation, sensations during the session, skin reactions, discomfort/adverse effects, and overall satisfaction. Items use ordered categorical response options (e.g., None/Mild/Moderate/Severe or Strongly disagree → Strongly agree), plus optional free-text. Outcome data will be reported as the number and proportion of participants in each response category for each item; free-text responses will be summarised narratively.
ABILHAND-Kids total raw score (0-42; higher = better manual ability) | Session 1[first visit]: Pre (Baseline, before tSCS); Session 1 [first visit]: Post (immediately after tSCS, within 10 minutes); Session 2 [second visit]: Pre (Baseline, before tSCS); Session 2 [sv]: Post (immediately after tSCS, within 10 minutes).
  Manual ability will be assessed with the ABILHAND-Kids Questionnaire (21 items; response options: Impossible = 0, Difficult = 1, Easy = 2). The total raw score is the sum across items (higher scores indicate better manual ability). The questionnaire may be completed by the participant or a caregiver proxy per instrument guidance. Results will be summarised as mean (SD) total score by timepoint and change from Pre to Post within each session (Post - Pre)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No